CLINICAL TRIAL: NCT05955859
Title: Diagnostics of Mycotic Sinusitis in Patients With Unilateral Obfuscation of the Paranasal Sinus and Patients With Uni-lateral Discharge From the Nasal Cavity
Brief Title: Diagnostics of Mycotic Sinusitis in ENT Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KORLCHHK-2023-Mycosis; 06-RVO-FNOs/2023 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fungal Sinusitis
Keywords: Sinusitis; Mycosis; Paranasal sinus
MeSH Terms: conditions — Sinusitis; Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with clinical suspicion of mycotic sinusitis (Experimental): Patient with clinical suspicion of mycotic sinusitis will undergo an examination as listed in Detailed Description.
  Interventions: Procedure: Samplings from patient's affected paranasal sinus

INTERVENTIONS:
Procedure: Samplings from patient's affected paranasal sinus — Samplings from patient's affected paranasal sinus during endoscopic surgery.

SUMMARY:
Mycotic sinusitis is a rare inflammatory disease of the paranasal sinuses. In recent years, its occurrence is increasing. Due to this situation, mycotic sinusitis is gaining importance, even though most cases of mycotic sinusitis are limited on paranasal sinuses.

Non-invasive forms of mycotic sinusitis are divided into mycetoma and allergic mycotic sinusitis. Mycetoma (fungus ball) usually affects only one paranasal sinus, most often maxillary sinus. The predisposing factors which participate on development of mycotic sinusitis are not exactly known. Some factors are considered as possible predisposing factors, for example deviation of nasal septum, dental treatment of upper jaw teeth or changes of nasal microbiome.

The diagnosis of fungal sinusitis is problematic. With the increasing number of patients, it is essential to improve the diagnostic process. In present, suspicion of mycotic sinusitis is based on the patient's clinical symptoms and the endoscopic findings in the nasal cavity. Only in some cases nonspecific findings can be observed, such as smelly secretions from the nose, feeling of stuffy nose and pain over the affected sinus. Some patients may be completely asymptomatic, and only in some cases fungal masses can be observed in the nasal cavity. Computed tomography (CT) scans are gaining more and more importance. Typical sign of an affected sinus is obfuscation on CT scan but this sign is not specific for mycotic infection. Central hyperdense foci are also present in some patients, but they are also not specific and can imitate a foreign body. Identifying specific signs on CT scan could help with diagnosing mycotic sinusitis.

DETAILED DESCRIPTION:
To identify specific determining signs for the diagnosis of fungal sinusitis, patients will undergo a series of examinations listed below.

1. Entrance ear, nose, throat (ENT) examination

   * anamnesis (nasal secretion, nasal obstruction, nose injury, dental procedures on the teeth of the upper jaw, immune disorder)
   * rhinological questionnaires (SNOT-22, rhinoVAS, NOSE score, olfactory questionnaire)
   * ENT examination without endoscope: deviation of the nasal septum or hypertrophy of the nasal conchae, pathological secretion from the nose
   * endoscopic examination of the nose: pathological secretion in the nasal cavity or from the orifice of the sinuses, the presence of fungal masses in the nasal cavity, obstruction of the orifice of the sinuses, the edge of the nasal septum
2. Computed tomography (CT) examination of the paranasal sinuses

   * evaluation of images in the frontal, sagittal and transverse planes
   * criteria of the affected cavity - complete/partial obscuration of the paranasal sinuses, hyperdense core, usuration or thickening of the bone of the paranasal sinuses
   * anatomical conditions of the nose and paranasal sinuses - the presence of septal deviation, dental pathology, Onodi's cellar, Haller's cellar, lateral recess of the sphenoid sinus
3. Functional endonasal endoscopic surgery (FESS)

   * method of execution performance of functional endonasal endoscopic surgery - only the affected cavity is being operated, complete cleaning of the affected cavity
   * sampling during surgery (4 in total): two samples for histological examination (sample 1 - mycotic material, sample 2 - mucous of the affected paranasal sinus), sample 3 - mycotic material for culture examination of fungi, sample 4 - mycotic material for elemental analysis using electron microscopy .
4. postoperative sample analysis

   * elemental analysis (sample 4): before analysis - control X-ray examination of the sample, the presence of hyperdense material on the X-ray image, performing electron microscopy, according to the structure of element evaluation.
   * histological examination (sample 1 and 2): evaluation of the sample 2 - mucosa of the paranasal sinuses - the presence of fungal invasion into the mucosa, inflammatory cellulization in the mucosa, evaluation of the sample 1 (mycotic material) - the presence of hyphae, inflammatory cellulization, calcification.
   * culture examination (sample 3): evaluation of the cultured finding by a microbiologist

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* patients with unilateral obfuscation of the paranasal sinus and patients with unilateral discharge from the nasal cavity

Exclusion Criteria:

* serious illness (decompensation phase) - cardiac, liver, kidney disease, can-cer
* serious psychiatric illnesses
* pregnancy
* high operative risk according to The American Society of Anesthesiologists (ASA) ≥ IV
* disagreement with participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Computer tomography (CT) examination of the paranasal sinuses - images | 3 years
  Evaluation of images in the frontal, sagittal and transverse planes - condition assessment.
Computer tomography (CT) examination of the paranasal sinuses - criteria | 3 years
  Evaluation of criteria of the affected cavity - complete/partial obscuration of the paranasal sinuses, hyperdense core, usuration or thickening of the bone of the paranasal sinuses.
Computer tomography (CT) examination of the paranasal sinuses - anatomical conditions of the nose and paranasal sinuses | 3 years
  Evaluation of anatomical conditions of the nose and paranasal sinuses - the presence of septal deviation, dental pathology, Onodi's cellar, Haller's cellar, lateral recess of the sphenoid sinus.
Entrance ENT examination - anamnesis | 3 years
  Taking anamnesis from patients to summarize any nasal secretion, nasal obstruction, nose injury, dental procedures on the teeth of the upper jaw or immune disorder.
Entrance ENT examination - SNOT-22 | 3 years
  Sino-Nasal Outcome Test-22 (SNOT-22) Questionnaire - The patients will complete a list of symptoms and social/emotional consequences of their nasal disorder. The SNOT-22 is a validated scale that measures sinonasal symptoms in patients with sinusitis. The 22 questions are scored on a scale of 0-5 with a maximum total score of 110. Higher scores represent more symptomatic patients.
Entrance ENT examination - rhinoVAS | 3 years
  Rhino Visual Analogue Scale (RhinoVAS) questionnaire will be used to assess postoperative changes in nasal function ranging from 0 (complete nose patency) to 10 cm (complete nose obstruction).
Entrance ENT examination - NOSE score | 3 years
  A simple, five-question, validated Nasal Obstruction Symptom Evaluation (NOSE) instrument that uses a 20-point scale to capture breathing symptoms, with higher scores indicating more severe symptoms than lower scores. A score of 0 means no problems with nasal obstruction and a score of 100 means the worst possible problems with nasal obstruction.
Entrance ENT examination - olfactory questionnaire | 3 years
  Olfactory questionnaire includes a short examination (test of identification and discrimination with perfumed markers) will be performed.
Entrance ENT examination - without endoscope | 3 years
  Observation of deviation of the nasal septum or hypertrophy of the nasal concha, patho-logical secretion from the nose.
Entrance ENT examination - endoscopic examination | 3 years
  Endoscopic examination of the nose in order to find any pathological secretion in the nasal cavity or from the orifice of the sinuses, the presence of fungal masses in the nasal cavity, obstruction of the orifice of the sinuses, the edge of the nasal septum.
Functional endonasal endoscopic surgery (FESS) - sample 1 | 3 years
  Mycotic material (as sample 1) for histological examination will be taken from patient´s affected cavity during FESS.
Functional endonasal endoscopic surgery (FESS) - sample 2 | 3 years
  Mucous of the affected paranasal sinus (as sample 2) for histological examination will be taken from patient´s affected cavity during FESS.
Functional endonasal endoscopic surgery (FESS) - sample 3 | 3 years
  Mycotic material for culture examination of fungi (as sample 3) will be taken from patient´s affected cavity during FESS.
Functional endonasal endoscopic surgery (FESS) - sample 4 | 3 years
  Mycotic material for elemental analysis using electron microscopy (as sample 4) will be taken from patient´s affected cavity during FESS.
Postoperative sample analysis - histological examination of sample 1 | 3 years
  Evaluation of the sample 1 (mycotic material) will be done to find out the presence of hyphae, inflammatory cellulization, calcification.
Postoperative sample analysis - histological examination of sample 2 | 3 years
  Evaluation of the sample 2 (mucosa of the paranasal sinuses) will be done to find out the presence of fungal invasion into the mucosa, inflammatory cellulization in the mucosa.
Postoperative sample analysis - culture examination of sample 3 | 3 years
  Evaluation of the cultured finding will be done by a microbiologist.
Postoperative sample analysis - elemental analysis of sample 4 | 3 years
  Control X-ray examination of the sample will be taken before analysis to find out the presence of hyperdense material on the X-ray image. Performing electron microscopy, according to the structure of ele-ment evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Polášková, MD, Principal Investigator — University Hospital Ostrava; Petr Matoušek, MD, Ph.D., Study Chair — University Hospital Ostrava; Michaela Masárová, MD, Study Chair — University Hospital Ostrava; Pavel Komínek, Prof., MD, Ph.D., Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Department of Otorhinolaryngology and Head and Neck Surgery, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.